CLINICAL TRIAL: NCT06065293
Title: Establishing a Community-led, Family-centered Mental Wellness Initiative in Rural Tanzania
Brief Title: Mental Health, Gender-Based Violence, and Stunting in Tanzania
Status: Completed | Type: Observational
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Other Study IDs: 3916
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Mental Health Issue; Substance Use; Child Development
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mothers involved in a local non-profit

SUMMARY:
One in three children under the age of five in Tanzania experience stunting, which is defined as impairments in growth and development that often occur after poor nutrition, poor health, and low psychosocial stimulation. Research suggests that mental health problems of parents may be related to stunting outcomes and parental mental health is closely related to experiences of intimate partner violence, also called gender-based violence. However, very little research exists on the connection between these elements, and interventions may be necessary in order to reduce the impacts that mental health and gender-based violence may have on stunting.

This study is a secondary data analysis of de-identified survey and stunting data that were conducted as a part of a needs assessment by a local nonprofit organization in Tanzania. The needs assessment was conducted to inform a mental health initiative organized by the established nonprofit across 5 villages in rural Tanzania. This project's primary aims are:

* To determine the prevalence of mental health and family relationship problems in five villages
* To determine associations between intimate partner violence (IPV) mental health and substance use and childhood stunting

ELIGIBILITY:
Inclusion Criteria:

* Living within the 5 rural villages
* participating in a local nonprofit
* pregnant or having a child under 2 years old

Exclusion Criteria:

* Living outside of the 5 villages
* Not participating in the local nonprofit
* Not pregnant or having a child under 2 years old

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 162 mothers participating in a local non-profit organization in Tanzania
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Depression and anxiety | Through study completion, approximately 2 months
  Hopkins Symptom Checklist
Substance use | Through study completion, approximately 2 months
  Alcohol Use Disorders Identification Test (AUDIT)
World Health Organization (WHO) Violence Against Women | Through study completion, approximately 2 months
  WHO Violence Against Women
Childhood stunting | Through study completion, approximately 2 months
  Height, weight, and head circumference of child under 2.5 years old

SECONDARY OUTCOMES:
Women's Empowerment | Through study completion, approximately 2 months
  Women's Empowerment measure

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Haddock, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The data are de-identified and there is no plan to make it available to other researchers